CLINICAL TRIAL: NCT03550222
Title: Muscle Evaluation Using Ultrasound in the Critically Ill : ULTRAMUSCLE Study
Brief Title: Muscle Evaluation Using Ultrasound in the Critically Ill
Acronym: ULTRAMUSCLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0302
Record Dates: First submitted 2017-09-26; First posted 2018-06-08 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness; ICU Acquired Weakness
Keywords: Diaphragmatic dysfunction; Mechanical Ventilation; ICU acquired weakness; Weaning; Skeletal muscles; Respiratory muscles
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critical illness is associated with ICU acquired weakness and diaphragmatic dysfunction.

Ultrasound can evaluate the muscle mass non invasively and provides the ability for a muscle follow up during and after the ICU stay. Magnetic stimulation of the phrenic nerves and the measure of the end expiratory tracheal pressure with an occlusion valve allows to evaluate the diaphragm force production in mechanically ventilated patients.

The aim of the present study is to constitute an image bank and to describe the muscle mass and function recovery in critically ill patients.

DETAILED DESCRIPTION:
Critical illness is associated with ICU acquired weakness and diaphragmatic dysfunction.

Ultrasound can evaluate the muscle mass non invasively and provides the ability for a muscle follow up during and after the ICU stay. Magnetic stimulation of the phrenic nerves and the measure of the end expiratory tracheal pressure with an occlusion valve allows to evaluate the diaphragm force production in mechanically ventilated patients.

The aim of the present study is to constitute an image bank and to describe the mass and function recovery in critically ill patients.

Ultrasound and clinical data will be collected and analysed during the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with at least one organ failure defined, organ failure being defined by a SOFA equal or above 3 for the organ, and an expected duration of ICU stay equal of above 3 days

Exclusion criteria:

- Pregnancy, age below 18, absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with at least one organ failure and an estimated duration of ICU stay of 3 days or more
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound characteristics of the quadriceps | Since admission at day 0 and measured repetitively by 48 hours untildischarge from ICU or date of death from any cause, whichever came first, assessed up to day 28
  Changes in ultrasound characteristics of the quadriceps : cross sectional area of quadriceps (cm2)

OTHER OUTCOMES:
Ultrasound characteristics of the biceps | Since admission at day 0 and measured repetitively by 48 hours untildischarge from ICU or date of death from any cause, whichever came first, assessed up to day 28
  Changes in ultrasound characteristics of the biceps : thickness of the biceps (mm)
Ultrasound characteristics of the diaphragm | Since admission at day 0 and measured repetitively by 48 hours untildischarge from ICU or date of death from any cause, whichever came first, assessed up to day 28
  Ultrasound characteristics of the diaphragm : thickness (mm)

CONTACTS AND LOCATIONS:
Overall Officials: BORIS JUNG, MD, PhD, Study Chair — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Aarab Y, Flatres A, Garnier F, Capdevila M, Raynaud F, Lacampagne A, Chapeau D, Klouche K, Etienne P, Jaber S, Molinari N, Gamon L, Matecki S, Jung B. Shear Wave Elastography, a New Tool for Diaphragmatic Qualitative Assessment: A Translational Study. Am J Respir Crit Care Med. 2021 Oct 1;204(7):797-806. doi: 10.1164/rccm.202011-4086OC. PMID 34255974
- [Derived] Flatres A, Aarab Y, Nougaret S, Garnier F, Larcher R, Amalric M, Klouche K, Etienne P, Subra G, Jaber S, Molinari N, Matecki S, Jung B. Real-time shear wave ultrasound elastography: a new tool for the evaluation of diaphragm and limb muscle stiffness in critically ill patients. Crit Care. 2020 Feb 3;24(1):34. doi: 10.1186/s13054-020-2745-6. PMID 32014005